CLINICAL TRIAL: NCT00952393
Title: Nicotinic Receptors and Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHBB-005-09S
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
Keywords: receptors nicotinic
MeSH Terms: conditions — Schizophrenia | interventions — Pharmacogenomic Variants; 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pharmacokinetic (Other): This single arm examines the pharmaco-kinetics of the release of 3-2,4 dimethoxy-benzilidene anabaseine in a hypomellose sustained release formulation.
  Interventions: Drug: Pharmacokinetic

INTERVENTIONS:
Drug: Pharmacokinetic — Subject receives 150 mg of compound formulated with hypomellose and Pharmcokinetics is determined
  Other Names: GTS-21

SUMMARY:
The study determines if a new preparation of a drug designed to treat schizophrenia is more slowly released into the body.

DETAILED DESCRIPTION:
3-2,4 dimethoxybenzylidene will be compounded with a methyallose compound in doses of 150 and 300 mg. The capsules will be administered singly and eventually bid to determine if sustained blood levels comparable to steady state blood levels seen in previous studies can be determined. Safety and EEG effects will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: males and females who are incapable of pregnancy

Exclusion Criteria:

* Medical illnesses requiring acute treatment
* History of seizures
* Substance abuse including nicotine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacokinetic
Started | 10 (10)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a collection of volunteers from the health science community who responded to approved advertisements.
Arm/Group | Pharmacokinetic
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years as determine by asking the subject when their birthdate is.
  years | 31.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants] — This is gender or sex as determined by inquiry from the subjects
  Participants
    Female | 3
    Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — We ask the subjects to report their ethnicity.
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 7
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — This is the area from which all the subjects come.
  participants
    United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Blood Levels of Drug
Description: This is the plasma level of the drug as determined by high performance liquid chromatography.
Time Frame: 12 hours
Population: This is all participants in the study.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Pharmacokinetic
Number analyzed (Participants) | 10
ng/ml | 1.5 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 24 hours.
Description: Subjects were questioned every hour for 8 hours and then 24 later, after administration of drug.
Arm/Group | Pharmacokinetic
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes